CLINICAL TRIAL: NCT04407702
Title: Control of Pain Due to Dentin Hypersensitivity in Individuals With Molar-incisor Hypomineralization: Study Protocol for a Randomized, Controlled, Clinical Trial
Brief Title: Control of Pain Due to Dentin Hypersensitivity in Individuals With Molar-incisor Hypomineralization
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hypersensitivity
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Dentin Sensitivity; Molar Incisor Hypomineralization
MeSH Terms: conditions — Dentin Sensitivity; Molar Hypomineralization | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All volunteers and the evaluator of the degree of sensitivity will be blinded to the allocation. The researcher in charge of applying the products will not be blinded due to the different forms of clinical manipulation of the products.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Experimental): The volunteers in this group will receive the same hygiene instructions as the other groups and will undergo both treatments, except that water will be used instead of the sealant and the laser device will be set to a power of 0 W. In other words, the same irradiation procedure will be performed but without the emission of light.
  Interventions: Other: Hygiene Instructions
- Sealant Group (Experimental): The volunteers in this group will receive treatment with sealant (Permaseal - Ultradent), which is a photopolymerizable methacrylate-based resin.
  Interventions: Other: Hygiene Instructions; Procedure: Sealant application
- Low-Level Laser Group (Experimental): The volunteers in this group will receive irradiation with AsGaAl laser at a wavelength of 780 nm (Laser XT Therapy, DMC, São Carlos, SP, Brazil) with relative isolation.
  Interventions: Other: Hygiene Instructions; Radiation: Low-level Laser
- Low Level Laser + Sealant Group (Experimental): The volunteers in this group will receive the same irradiation administered to Low-level Laser Group. During the last session, these volunteers will also receive the same sealant applied in Sealant Group.
  Interventions: Other: Hygiene Instructions; Procedure: Sealant application; Radiation: Low-level Laser

INTERVENTIONS:
Other: Hygiene Instructions — Two weeks prior to the onset of the study, the volunteers will undergo a wash-out period, in which they will only use oral hygiene products donated by the researchers. These products will be used through to the end of the study. The oral hygiene kit will contain a soft-bristle toothbrush (Professional Lab Series, Colgate Palmolive), fluoride toothpaste with no desensitizing agent (Elmex) and dental floss (Colgate). The participants will be extensively trained with regards to all procedures involved in the experiment.
Procedure: Sealant application — The teeth to be sealed will be isolated and 35% phosphoric acid will be applied for 20 seconds, followed by rinsing and drying the dental surfaces. A thin layer of PermaSeal will be applied to the tooth surface for 5 seconds and photopolymerized for 20 seconds. The occlusion will then be evaluated.
  Arms: Low Level Laser + Sealant Group; Sealant Group
Radiation: Low-level Laser — Irradiation with AsGaAl laser at a wavelength of 780 nm (Laser XT Therapy, DMC, São Carlos, SP, Brazil) with relative isolation. The power will be set to 100 mW; energy density will be 35 J/cm2 (considering a spot size of 0.028 cm2 of the equipment) and the dose will be 1 J per point. Irradiation will be performed on a cervical point, an apical point and a point precisely over the lesion, totaling a dose of 3 J. Treatment will be performed in three sessions with a 72-hour interval between sessions.
  Arms: Low Level Laser + Sealant Group; Low-Level Laser Group

SUMMARY:
Background: Dentin hypersensitivity (DH) is defined as high sensitivity of the vital dentin when exposed to thermal, chemical or tactile stimuli. Two mechanisms are required for the occurrence of DH: 1) the dentin must be exposed and 2) the dentinal tubules must be open and connected to the pulp. Molar-incisor hypomineralization (MIH) is a qualitative abnormality of a genetic origin that affects tooth enamel and, in most cases, is accompanied by DH. The control of tooth sensitivity is fundamental to the successful treatment of MIH.

Objective: The aim of the proposed randomized, controlled, clinical trial is to evaluate the effectiveness of different protocols for the control of DH in patients with teeth affected by MIH.

Methods: One hundred forty patients who meet the inclusion criteria will be allocated to four groups. Group 1 will be the control group (placebo). In Group 2, sensitive teeth will be sealed with Permaseal (Ultradent). In Group 3, sensitive teeth will receive low-level laser (LLL) (AsGaAl) at a wavelength of 780 nm (Laser XT Therapy, DMC, São Carlos, SP, Brazil). In Group 4, sensitive teeth will be treated with both LLL and Permaseal (Ultradent). DH will be evaluated 15 min after the application of the treatments and the patients will be reevaluated one week, one month, three months and six months after the treatments.

Discussion: This study will enable the determination of differences in the effectiveness of the proposed treatments as well as differences among the evaluation times for each proposed treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years;
* Good overall health;
* At least one tooth with MIH and DH reported in the cervical region with sensitivity equal to or greater than 4 on the VAS.

Exclusion Criteria:

* Active caries or defective restorations on the tooth to be analyzed;
* Sufficient dentin loss that requires restorative treatment or periodontal surgery;
* Having undergone any professional desensitizing treatment in the previous six months;
* Having used a desensitizing paste in the previous three months;
* Use of anti-inflammatory drugs or analgesics at the time of recruitment;
* Currently pregnant or nursing.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
Change in pain evaluated through a Visual Analog Scale (VAS) | Baseline, one week, one month, three months and six months after the final treatment session.
  The researcher will assess the sensitive tooth using cold air from the triple syringe (2 s of compressed air at a pressure of approximately 40 psi with the syringe perpendicular to the tooth surface at a distance of approximately 0.5 cm). Neighboring teeth will be protected with cotton rolls or the examiner's fingers9. The volunteer will then indicate a whole number between 0 (absence of pain) to 10 (worst pain possible) on the 10-cm VAS scale that best describes his/her perception of pain.

IPD SHARING:
Plan to Share IPD: Yes
The datasets (Excel spreadsheets) generated from this protocol will be available with the corresponding author (Sandra Kalil Bussadori - sandra.skb@gmail.com) at a reasonable request. However, reuse of this data will not be allowed for people who are not authors of this paper.

REFERENCES:
- [Derived] Sobral APT, Santos EM, Aranha AC, Soares PV, Moriyama CM, Goncalves MLL, Ribeiro RA, Motta LJ, Horliana ACRT, Fernandes KPS, Mesquita-Ferrari RA, Bussadori SK. The control of pain due to dentin hypersensitivity in individuals with molar-incisor hypomineralisation: a protocol for a randomised controlled clinical trial. BMJ Open. 2021 Mar 10;11(3):e044653. doi: 10.1136/bmjopen-2020-044653. PMID 33692185